CLINICAL TRIAL: NCT02004652
Title: A Randomized, Controlled, Double-blind Efficacy and Tolerability Study Of Prucalopride For The Treatment Of Postoperative Ileus In Patients Undergoing Gastrointestinal Surgery
Brief Title: Prucalopride for Postoperative Ileus in Patients Undergoing Gastrointestinal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIGS-2013-PRU
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Ileus
Keywords: Prucalopride; Gastrointestinal Diseases; Postoperative ileus; Randomised trial
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prucalopride (Experimental): Prucalopride, 2mg, tablet. First given 24 hours after surgery beginning on POD 1,until bowel movements or for a maximum of 7 days of postoperative treatment
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator): Vitamin C, 50mg, tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — Prucalopride, 2mg, tablet. First given 24 hours after surgery beginning on POD 1,until bowel movements or for a maximum of 7 days of postoperative treatment
  Other Names: Resolor
  Arms: Prucalopride
Drug: Placebo — Vitamin, 50mg, tablet.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect and safety of prucalopride on recovery of gastrointestinal function in patient undergoing major gastrointestinal surgery. The investigators hypothesize that patients who take prucalopride after major gastrointestinal surgery will have shorter duration of postoperative ileus.

DETAILED DESCRIPTION:
Postoperative ileus (POI), an interruption of bowel motility function, virtually occurs in all patients undergoing major gastrointestinal(GI) surgery. This functional impairment persists for a variable duration, usually resolving within 1 day in the small intestine, 1 to 3 days in the stomach and 3 to 5 days in the colon. Therefore, time of return of colonic function is the the major determinant of duration of POI. Attempts to reduce the duration of POI have prompted the implementation of fast track surgery including early removal of the nasogastric tube, early feeding, alvimopan, gum chewing, and prompt ambulation. However, it is still reported to be more than 4-5 days in most of the randomized trial. Therefore, methods specifically aiming at promoting postoperative colon motility may further enhance the GI function recovery, and prucalopride may be one of the options.

Prucalopride, a substituted benzamide with selective 5-HT4 agonist activity, has been shown previously to significant improve colon motility and transit, but it only has mild effect on gastric or small bowel transit. The drug is well tolerated with no significant adverse effects. Recently, prucalopride has been approved in Europe and America for the symptomatic treatment of chronic constipation in women in whom laxatives fail to provide adequate relief. However, its usage in the postoperative period has not been tested. This study will test the ability and safety of prucalopride given 24hrs after GI surgery to hasten the recovery of GI function.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients undergoing elective gastric, small bowel, or partial colonic resection via laparotomy or laparoscopy.
2. Patients with American Society of Anaesthesiologists grading I-III
3. Informed consent available.

Exclusion Criteria:

1. Patients with stoma creation, extensive adhesiolysis, total or subtotal colectomy , or patients who had a history of total or subtotal colectomy.
2. Patients who developed intraoperative problems or complications, or had peritoneal carcinomatosis.
3. Patients who developed serious complications within 24 hours after surgery.
4. Those who received epidural anesthesia or analgesia.
5. Patients who received other prokinetic drugs.
6. Patients who were allergic to prucalopride.
7. Patients with severe comorbidity and/or organ(kidney, liver, and heart) dysfunction
8. Patients had complete bowel obstruction
9. Patients who have participated other clinical trials.
10. Patients who have short bowel(<200cm small bowel) or history of constipation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to defaecation, measured in hours, from the time the surgery ends till the first observed passage of stool | up to 30 days after surgery

SECONDARY OUTCOMES:
Time of first passing flatus reported by the patients(hours) | up to 30 days after surgery
Time to resume solid diet or total enteral nutrition(TEN)(days) | up to 30 days after surgery
Length of postoperative hospital stay (LOS)(days) | participants will be followed for the duration of postoperative hospital stay, an expected average of 8 days
Overall post-operative complication rate defined according to the Clavien-Dindo Classification | up to 30 days after surgery
Overall cost (RMB) | participants will be followed for the duration of postoperative hospital stay, an expected average of 8 days
Pain scores on visual analogue scale (from 0 which implies no pain at all, to 10 which implies the worst pain imaginable) on the first 3 postoperative days and postoperative analgesic requirement (number of doses on 50-mg Pethidine) | up to postoperative day 3
Time to walk independently(days) | up to 30 days after surgery
Hospital Readmission Rates Post 30-day Discharge | up to 30 days after discharge
Length of postoperative ICU stay (days) | up to 30 days after surgery
Incidence of adverse events related to drug usage | up to 7 days after drug usage
  Diarrhoea,Flatulence,Nausea,Abdominal pain,Headaches,Menstrual disorder,Dizziness ,Skeletal pain,ECG nodal arrhythmia
Reinsertion of nasogastric tube | up to 30 days after surgery

OTHER OUTCOMES:
Whole blood white blood cell(WBC) count on postoperative day 1 and 3 | postoperative day 1 and 3
  whole blood white blood cell (WBC) count(*109/L)
Whole blood neutrophil percentage on postoperative day 1 and 3 | postoperative day 1 and 3
  neutrophil percentage(%)
Whole blood platelet level on postoperative day 1 and 3 | postoperative day 1 and 3
  platelet level(*109/L)
Serum C-reactive protein(CRP) level on postoperative day 1 and 3. | postoperative day 1 and 3
  CRP level(mg/dL)
Serum interleukin-6(IL-6) level on postoperative day 1 and 3. | postoperative day 1 and 3
  IL-6(pg/ml)
Serum procalcitonin(PCT) level on postoperative day 1 and 3. | postoperative day 1 and 3
  PCT(ug/L)

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Gong, MD, Principal Investigator — Department of general surgery,Jinling hospital
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Gong J, Xie Z, Zhang T, Gu L, Yao W, Guo Z, Li Y, Lu N, Zhu W, Li N, Li J. Randomised clinical trial: prucalopride, a colonic pro-motility agent, reduces the duration of post-operative ileus after elective gastrointestinal surgery. Aliment Pharmacol Ther. 2016 Apr;43(7):778-89. doi: 10.1111/apt.13557. Epub 2016 Feb 15. PMID 26880227